CLINICAL TRIAL: NCT00804687
Title: A Randomized, Single-Dose, Single-Blind, Double-Dummy, Placebo-Controlled, Three-Way Cross-Over Study to Compare the Relative Efficacy of JNJ-39220675, Pseudoephedrine and Placebo for the Treatment of Allergic Rhinitis in an Environmental Exposure Chamber (EEC) Model
Brief Title: An Efficacy Study of JNJ-39220675 and Pseudoephedrine in Participants With Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR015709; 39220675ATT2001
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Allergic Rhinitis
Keywords: Allergy; Rhinitis; Allergic Rhinitis; JNJ-39220675; Pseudoephedrine
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity; Rhinitis | interventions — (4-cyclobutyl-(1,4)diazepan-1-yl)-(6-(4-fluorophenoxy)pyridin-3-yl)methanone; Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- JNJ-39220675 then Pseudoephedrine then Placebo (Experimental): Single-dose of JNJ-39220675 will be administered as 1 milliliter (ml) of 10 milligram/milliliter (mg/ml) solution orally along with placebo tablet in first treatment period; after that in second treatment period, single-dose of 1 ml placebo solution will be administered orally along with 60 milligram (mg) pseudoephedrine tablet; and then single-dose of 1 ml placebo solution will be administered orally along with placebo tablet in third treatment period. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Other: Placebo; Drug: JNJ-39220675; Drug: Pseudoephedrine
- JNJ-39220675 then Placebo then Pseudoephedrine (Experimental): Single-dose of JNJ-39220675 will be administered as 1 ml of 10 mg/ml solution orally along with placebo tablet in first treatment period; after that, in second treatment period, single-dose of 1 ml placebo solution will be administered orally along with placebo tablet; and then single-dose of 1 ml placebo solution will be administered orally along with 60 mg pseudoephedrine tablet in third treatment period. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Other: Placebo; Drug: JNJ-39220675; Drug: Pseudoephedrine
- Placebo then JNJ-39220675 then Pseudoephedrine (Experimental): Single-dose of 1 ml placebo solution will be administered orally along with placebo tablet in first treatment period; after that, in second treatment period, single-dose of JNJ-39220675 will be administered as 1 ml of 10 mg/ml solution orally along with placebo tablet; and then single-dose of 1 ml placebo solution will be administered orally along with 60 mg pseudoephedrine tablet in third treatment period. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Other: Placebo; Drug: JNJ-39220675; Drug: Pseudoephedrine
- Placebo then Pseudoephedrine then JNJ-39220675 (Experimental): Single-dose of 1 ml placebo solution will be administered orally along with placebo tablet in first treatment period; after that, in second treatment period, single-dose of 1 ml placebo solution will be administered orally along with 60 mg pseudoephedrine tablet; and then single-dose of JNJ-39220675 will be administered as 1 ml of 10 mg/ml solution orally along with placebo tablet in third treatment period. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Other: Placebo; Drug: JNJ-39220675; Drug: Pseudoephedrine
- Pseudoephedrine then JNJ-39220675 then Placebo (Experimental): Single-dose of 1 ml placebo solution will be administered orally along with 60 mg pseudoephedrine tablet in first treatment period; after that, in second treatment period, single-dose of JNJ-39220675 will be administered as 1 ml of 10 mg/ml solution along with placebo tablet; and then single-dose of 1 ml placebo solution will be administered orally along with placebo tablet in third treatment period. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Other: Placebo; Drug: JNJ-39220675; Drug: Pseudoephedrine
- Pseudoephedrine then Placebo then JNJ-39220675 (Experimental): Single-dose of 1 ml placebo solution will be administered orally along with 60 mg pseudoephedrine tablet in first treatment period; after that, in second treatment period, single-dose of 1 ml placebo solution will be administered orally along with placebo tablet; and then single-dose of JNJ-39220675 will be administered as 1 ml of 10 mg/ml solution orally along with placebo tablet in third treatment period. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Other: Placebo; Drug: JNJ-39220675; Drug: Pseudoephedrine

INTERVENTIONS:
Other: Placebo — Single-dose of 1 milliliter (ml) placebo solution will be administered orally and/or placebo tablet orally in one of the treatment periods.
Drug: JNJ-39220675 — Single-dose of JNJ-39220675 will be administered as 1 ml of 10 milligram/milliliter solution orally in one of the treatment periods.
Drug: Pseudoephedrine — Single-dose of 60 milligram pseudoephedrine tablet will be administered orally in one of the treatment periods.

SUMMARY:
The purpose of this study is to evaluate the relative efficacy of JNJ- 39220675 and pseudoephedrine compared to placebo (medication with no active ingredients) in participants with allergic rhinitis (inflammation of the nose due to exposure to allergens such as pollen, dust or animal hair).

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), single-dose, single-blind (a clinical trial in which the person giving the treatment, but not the participant, knows which treatment the participant is receiving), double-dummy, placebo-controlled, three-treatment period, cross-over (participants may receive different interventions sequentially during the trial) study of JNJ-39220675 in participants with allergic rhinitis. The duration of study will be 20-64 days per participant. The study consists of 2 parts: Screening (that is, 30 days before study commences on Day 1) and Treatment (consists of single-dose of either JNJ-39220675 solution [10 milligram], Pseudoephedrine tablet [60 milligram] or Placebo, in subsequent three-treatment periods, each separated with washout period of 6 days). All the eligible participants will be randomly assigned to 1 of the 6 treatment sequences. Participants will be given dose approximately 2 hours before entry into the environmental exposure chamber where they will be exposed to ragweed pollen for 8 hours. Efficacy will primarily be evaluated by measurement of nasal congestion that will be assessed through nasal cavity geometry that is, minimal cross-sectional area of nasal cavity by Acoustic rhinometry. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a clinical history of seasonal allergic rhinitis with seasonal onset and offset of nasal allergy symptoms at least during each of the last two ragweed allergy seasons
* Participants must have documentation of a positive skin test within 12 months of Screening to ragweed allergen defined by a positive case history and a positive skin prick and/or intradermal test (allergy tests performed by injecting allergy-causing substances underneath the skin to see if they cause a reaction) for ragweed allergen
* Female participants must not be pregnant, lactating or be able to become pregnant
* Male participants must consent to use a medically acceptable method of contraception throughout the entire study period and for 3 months after the study is completed
* Participants with body mass index between 18 and 32 kilogram per square meter

Exclusion Criteria:

* Participants with clinically significant physical findings of nasal anatomical deformities
* Participants with a history of risk factors for torsades de pointes (heart failure, hypokalemia, family history of long QT syndrome), use of concomitant medications that prolong the QT or QTc interval or an abnormal 12-lead electrocardiogram except for clinically non-significant bradycardia
* Participants with history of exposure to an investigational treatment within the 30 days before the Screening Visit, or has ever taken JNJ-39220675 previously
* Participants with a history of clinically significant allergies, especially known hypersensitivity or intolerance to any drug or known allergy to the study drug or any of the excipients of the formulation
* Participants with a history of severe respiratory infection or disorder, epilepsy or seizures, coronary heart disease, uncontrolled hypertension, or other clinically significant cardiovascular disease, or history of a positive test for Human immuno-deficiency (HIV), Hepatitis B or Hepatitis C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- JNJ-39220675 Then Pseudoephedrine Then Placebo: Single-dose of JNJ-39220675 as 1 milliliter (ml) of 10 milligram/milliliter (mg/ml) solution orally and placebo tablet orally in first treatment period; after that single-dose of 1 ml placebo solution orally and 60 milligram (mg) pseudoephedrine tablet orally in second treatment period; and then single-dose of 1 ml placebo solution orally and placebo tablet orally in third treatment period. A washout period of at least 6 days was maintained between each treatment period.
- JNJ-39220675 Then Placebo Then Pseudoephedrine: Single-dose of JNJ-39220675 as 1 ml of 10 mg/ml solution orally and placebo tablet orally in first treatment period; after that single-dose of 1 ml placebo solution orally and placebo tablet orally in second treatment period; and then single-dose of 1 ml placebo solution orally and 60 mg pseudoephedrine tablet orally in third treatment period. A washout period of at least 6 days was maintained between each treatment period.
- Placebo Then JNJ-39220675 Then Pseudoephedrine: Single-dose of 1 ml placebo solution orally and placebo tablet orally in first treatment period; after that single-dose of JNJ-39220675 as 1 ml of 10 mg/ml solution orally and placebo tablet orally in second treatment period; and then single-dose of 1 ml placebo solution orally and 60 mg pseudoephedrine tablet orally in third treatment period. A washout period of at least 6 days was maintained between each treatment period.
- Placebo Then Pseudoephedrine Then JNJ-39220675: Single-dose of 1 ml placebo solution orally and placebo tablet orally in first treatment period; after that single-dose of 1 ml placebo solution orally and 60 mg pseudoephedrine tablet orally in second treatment period; and then single-dose of JNJ-39220675 as 1 ml of 10 mg/ml solution orally and placebo tablet orally in third treatment period. A washout period of at least 6 days was maintained between each treatment period.
- Pseudoephedrine Then JNJ-39220675 Then Placebo: Single-dose of 1 ml placebo solution orally and 60 mg pseudoephedrine tablet orally in first treatment period; after that single-dose of JNJ-39220675 as 1 ml of 10 mg/ml solution orally and placebo tablet orally in second treatment period; and then single-dose of 1 ml placebo solution orally and placebo tablet orally in third treatment period. A washout period of at least 6 days was maintained between each treatment period.
- Pseudoephedrine Then Placebo Then JNJ-39220675: Single-dose of 1 ml placebo solution orally and 60 mg pseudoephedrine tablet orally in first treatment period; after that single-dose of 1 ml placebo solution orally and placebo tablet orally in second treatment period; and then single-dose of JNJ-39220675 as 1 ml of 10 mg/ml solution orally and placebo tablet orally in third treatment period. A washout period of at least 6 days was maintained between each treatment period.
Period: Period 1: Treatment Period
Arm/Group | JNJ-39220675 Then Pseudoephedrine Then Placebo | JNJ-39220675 Then Placebo Then Pseudoephedrine | Placebo Then JNJ-39220675 Then Pseudoephedrine | Placebo Then Pseudoephedrine Then JNJ-39220675 | Pseudoephedrine Then JNJ-39220675 Then Placebo | Pseudoephedrine Then Placebo Then JNJ-39220675
Started | 9 | 9 | 9 | 9 | 9 | 8
Completed | 9 | 9 | 9 | 9 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2: Washout Period
Arm/Group | JNJ-39220675 Then Pseudoephedrine Then Placebo | JNJ-39220675 Then Placebo Then Pseudoephedrine | Placebo Then JNJ-39220675 Then Pseudoephedrine | Placebo Then Pseudoephedrine Then JNJ-39220675 | Pseudoephedrine Then JNJ-39220675 Then Placebo | Pseudoephedrine Then Placebo Then JNJ-39220675
Started | 9 | 9 | 9 | 9 | 9 | 8
Completed | 9 | 9 | 9 | 9 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3: Treatment Period
Arm/Group | JNJ-39220675 Then Pseudoephedrine Then Placebo | JNJ-39220675 Then Placebo Then Pseudoephedrine | Placebo Then JNJ-39220675 Then Pseudoephedrine | Placebo Then Pseudoephedrine Then JNJ-39220675 | Pseudoephedrine Then JNJ-39220675 Then Placebo | Pseudoephedrine Then Placebo Then JNJ-39220675
Started | 9 | 9 | 9 | 9 | 9 | 8
Completed | 9 | 9 | 9 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Positive Drug screen | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 4: Washout Period
Arm/Group | JNJ-39220675 Then Pseudoephedrine Then Placebo | JNJ-39220675 Then Placebo Then Pseudoephedrine | Placebo Then JNJ-39220675 Then Pseudoephedrine | Placebo Then Pseudoephedrine Then JNJ-39220675 | Pseudoephedrine Then JNJ-39220675 Then Placebo | Pseudoephedrine Then Placebo Then JNJ-39220675
Started | 9 | 9 | 9 | 8 | 9 | 8
Completed | 9 | 9 | 9 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5: Treatment Period
Arm/Group | JNJ-39220675 Then Pseudoephedrine Then Placebo | JNJ-39220675 Then Placebo Then Pseudoephedrine | Placebo Then JNJ-39220675 Then Pseudoephedrine | Placebo Then Pseudoephedrine Then JNJ-39220675 | Pseudoephedrine Then JNJ-39220675 Then Placebo | Pseudoephedrine Then Placebo Then JNJ-39220675
Started | 9 | 9 | 9 | 8 | 9 | 8
Completed | 8 | 9 | 8 | 8 | 8 | 8
Not Completed | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Positive drugs of abuse | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Positive drug test | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants randomized in the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 53
Age Continuous [Mean (Standard Deviation); unit: years] | 41.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Baseline Adjusted Area Under the Curve (AUC) of Minimal Cross-Sectional Area (MCA) of Nasal Cavity by Acoustic Rhinometry
Description: The AcR was an objective measurement of nasal congestion that assessed nasal cavity geometry (that is, MCA) and changes in dimensions of nasal cavity. The AUC of MCA was used as response variable to assess treatment effect. AUC was adjusted for Baseline MCA scores. Baseline MCA was defined as minimum mean MCA at pre-dose (approximately 2 hours before Environmental Exposure Chamber [EEC] entry) resulting from 3 measurements on both, left and right nostrils in each of the treatment periods. The AUC of MCA was baseline-adjusted, by subtracting the Baseline value from each of the post-treatment times before calculating the AUC.
Time Frame: 2 and 0.5 hour before drug administration and 1, 2, 3, 4, 5, 6, 7 and 8 hours after drug administration at Day 1 of each treatment period
Population: Intent to treat (ITT) population included all participants who received at least one dose of study medication and had at least one post-baseline AcR efficacy assessment. 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: square centimeter*hour (cm^2*h)
Groups:
- Placebo: Single-dose of 1 milliliter placebo solution orally and/or placebo tablet orally in one of the treatment periods.
- JNJ-39220675: Single-dose of JNJ-39220675 as 1 ml of 10 milligram/milliliter solution orally in one of the treatment periods.
- Pseudoephedrine: Single-dose of 60 milligram pseudoephedrine tablet orally in one of the treatment periods.
Arm/Group | Placebo | JNJ-39220675 | Pseudoephedrine
Number analyzed (Participants) | 51 | 52 | 51
square centimeter*hour (cm^2*h) | -0.682 (0.803) | -0.504 (0.805) | -0.550 (0.843)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39220675; Test type: Superiority or Other; p = 0.0602, Linear mixed model; Least Squares Mean difference = -0.126, 95% CI [-0.258 to 0.006], Standard Error of Mean 0.066
Statistical Analysis 2: Comparison: Placebo vs Pseudoephedrine; Test type: Superiority or Other; p = 0.0043, Linear mixed model; Least Squares Mean difference = -0.195, 95% CI [-0.328 to -0.063], Standard Error of Mean 0.067
Statistical Analysis 3: Comparison: JNJ-39220675 vs Pseudoephedrine; Test type: Superiority or Other; p = 0.3513, Linear mixed model; Least Squares Mean difference = -0.066, 95% CI 2-sided [-0.206 to 0.075], Standard Error of Mean 0.070

2. Secondary Outcome: Baseline Adjusted Area Under the Curve (AUC) of Total Nasal Symptom Score (TNSS)
Description: The TNSS was the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Participants assessed each individual symptoms on a scale of 0-3 where: 0=absent, 1=mild, 2=moderate and 3=severe. TNSS score ranges from 0 to 12 and higher scores indicate worsening. The AUC of TNSS was used as response variable to assess the treatment effect. AUC was adjusted for Baseline TNSS scores. Baseline TNSS was defined as the symptom scores for each treatment period at pre-dose (approximately 2 hour before EEC entry).
Time Frame: 2, 1.5, 1, 0.5 hour before drug administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5 and 8 hours after drug administration at Day 1 of each treatment period
Population: The ITT population included all participants who received at least one dose of study medication and had at least one post-baseline AcR efficacy assessment. 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale * hours
Arm/Group | Placebo | JNJ-39220675 | Pseudoephedrine
Number analyzed (Participants) | 51 | 52 | 51
units on a scale * hours | 45.720 (24.707) | 36.536 (24.322) | 43.195 (26.202)
Statistical Analysis 1: Comparison: Placebo vs JNJ-39220675; Test type: Superiority or Other; p = 0.0003, Linear mixed model; Least Squares Mean difference = 8.604, 95% CI [4.104 to 13.104], Standard Error of Mean 2.267
Statistical Analysis 2: Comparison: Placebo vs Pseudoephedrine; Test type: Superiority or Other; p = 0.0428, Linear mixed model; Least Squares Mean difference = 4.699, 95% CI [0.155 to 9.243], Standard Error of Mean 2.289
Statistical Analysis 3: Comparison: JNJ-39220675 vs Pseudoephedrine; Test type: Superiority or Other; p = 0.0895, Linear mixed model; Least Squares Mean difference = -3.905, 95% CI 2-sided [-8.424 to 0.614], Standard Error of Mean 2.277

3. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5 and 8 Hours After Drug Administration at Day 1
Description: The TNSS was the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Participants assessed each individual symptoms on a scale of 0-3 where: 0=absent, 1=mild, 2=moderate and 3=severe. TNSS score ranges from 0 to 12 and higher scores indicate worsening. Change from Baseline in TNSS is the value at particular time point minus value at Baseline.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5 and 8 hours after drug administration at Day 1 of each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-39220675 | Pseudoephedrine
Number analyzed (Participants) | 51 | 52 | 51
units on a scale
  Change at Hour 0.5 | 2.7 (3.0) | 1.4 (2.5) | 1.7 (2.4)
  Change at Hour 1 | 3.5 (3.5) | 2.2 (2.9) | 3.4 (3.6)
  Change at Hour 1.5 | 4.1 (3.8) | 3.2 (3.3) | 4.2 (3.7)
  Change at Hour 2 | 5.0 (3.6) | 3.9 (3.5) | 4.6 (3.8)
  Change at Hour 2.5 | 5.6 (3.7) | 4.1 (3.3) | 5.0 (3.7)
  Change at Hour 3.0 | 5.8 (3.6) | 4.7 (3.5) | 5.4 (3.5)
  Change at Hour 3.5 | 5.6 (3.5) | 4.9 (3.5) | 5.6 (3.6)
  Change at Hour 4 | 6.1 (3.6) | 5.4 (3.3) | 6.0 (3.8)
  Change at Hour 4.5 | 6.4 (3.4) | 5.3 (3.8) | 5.6 (3.8)
  Change at Hour 5 | 6.5 (3.4) | 5.3 (3.7) | 6.3 (3.6)
  Change at Hour 5.5 | 6.6 (3.2) | 5.4 (3.6) | 6.4 (3.7)
  Change at Hour 6 | 6.9 (3.5) | 5.6 (3.5) | 6.5 (3.6)
  Change at Hour 6.5 | 7.0 (3.4) | 5.7 (3.5) | 6.8 (3.8)
  Change at Hour 7 | 7.0 (3.5) | 6.1 (3.5) | 6.9 (3.7)
  Change at Hour 7.5 | 7.0 (3.6) | 6.1 (3.3) | 6.9 (3.5)
  Change at Hour 8 | 7.4 (3.4) | 6.5 (3.3) | 7.0 (3.6)

4. Secondary Outcome: Change From Baseline in Minimal Cross-Sectional Area (MCA) at 1, 2, 3, 4, 5, 6, 7 and 8 Hours After Drug Administration at Day 1
Description: The MCA was measured using AcR which is an objective measurement of nasal congestion that assesses nasal cavity geometry (that is, MCA) and changes in the dimensions of the nasal cavity. Change from Baseline in MCA is the value at particular time point minus value at Baseline.
Time Frame: Baseline, 1, 2, 3, 4, 5, 6, 7 and 8 hours after drug administration at Day 1 of each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: square centimeter (cm^2)
Arm/Group | Placebo | JNJ-39220675 | Pseudoephedrine
Number analyzed (Participants) | 51 | 52 | 51
square centimeter (cm^2)
  Baseline | 0.304 (0.106) | 0.294 (0.121) | 0.312 (0.116)
  Change at Hour 1 | -0.054 (0.112) | -0.028 (0.118) | -0.035 (0.118)
  Change at Hour 2 | -0.048 (0.122) | -0.041 (0.112) | 0.060 (0.111)
  Change at Hour 3 | -0.086 (0.114) | -0.055 (0.117) | -0.053 (0.115)
  Change at Hour 4 | -0.100 (0.105) | -0.077 (0.125) | -0.072 (0.119)
  Change at Hour 5 | -0.104 (0.124) | -0.082 (0.105) | -0.092 (0.127)
  Change at Hour 6 | -0.108 (0.117) | -0.091 (0.116) | -0.081 (0.148)
  Change at Hour 7 | -0.094 (0.135) | -0.079 (0.125) | -0.099 (0.124)
  Change at Hour 8 | -0.111 (0.119) | -0.090 (0.139) | -0.110 (0.115)

ADVERSE EVENTS:
Time Frame: Baseline up to End of Treatment (Day 41)
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable and unintended sign/abnormal finding, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Placebo | JNJ-39220675 | Pseudoephedrine
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 1/51 | 37/52 | 3/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | JNJ-39220675 (N=52) | Pseudoephedrine (N=51)
Palpitations (Cardiac disorders) | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 1 | 0
Mydriasis (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 7 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 5 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 9 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days